CLINICAL TRIAL: NCT07316127
Title: A Placebo-Controlled, Double-Blind, Randomized Trial Phase I-II With Immunoadsorption in Autoimmune Long COVID
Brief Title: Immunoadsorption in Autoimmune Long COVID
Acronym: TURNLongCOVID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, W. J. Wiersinga, MD, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL-009359
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Long COVID; Long COVID Syndrome; Long COVID-19 Syndrome; Post COVID Syndrome
Keywords: immunoadsorption; long COVID; post COVID; plasmapheresis
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Plasmapheresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Sham Comparator): Participants in the placebo group will receive six sessions of sham treament, each lasting 2.5 hours over two weeks. The procedure will be performed without an adsorption column, allowing the blood to circulate through the extracorporeal circuit and be returned to the patient without removal of immunoglobulins or other plasma components.
  Interventions: Device: Sham Comparator
- Immunoadsorption (Active Comparator): Participants in the intervention group will receive six sessions of immunoadsorption, each lasting 2.5 hours over two weeks. Immunoadsorption will be performed using tryptophan columns, which bind the Fc region of IgG via hydrophobic and aromatic interactions.
  Interventions: Device: Immunoadsorption

INTERVENTIONS:
Device: Immunoadsorption — Immunoadsorption will be performed using tryptophan columns, which bind the Fc region of IgG via hydrophobic and aromatic interactions.
  Arms: Immunoadsorption
Device: Sham Comparator — The immunoadsorption column will be removed from the device, so that the patient's blood passes through the system and is returned to the body without undergoing adsorption or removal of antibodies.
  Arms: Placebo

SUMMARY:
Some people continue to have serious symptoms long after COVID-19, such as extreme fatigue and feeling worse after activity. In some patients, this may happen because the immune system is attacking the body by mistake.

This study will test a treatment called immunoadsorption, which filters the blood to remove harmful antibodies. People with long COVID who have these antibodies will be randomly assigned to receive either the real treatment or a placebo. The main goal is to see whether fatigue improves after one month, and whether other symptoms and daily functioning improve over six months.

This research will help us find out if this treatment can benefit the group of long COVID patients with immune-related disease.

DETAILED DESCRIPTION:
Growing evidence indicates that autoantibodies may drive symptoms in a subset of people with long COVID, as demonstrated by symptom transfer to mice following administration of IgG from affected patients. This provides a strong rationale for targeted immunotherapy aimed at removing pathogenic antibodies. Immunoadsorption is a well-established method to reduce circulating IgG, but studies suggest that only a specific subgroup of patients benefits.

Using HuProt autoantibody microarray technology, we identified several autoantibodies uniquely present in long COVID patients compared with healthy controls. We subsequently developed and validated a disease-specific Luminex multiplex immunoassay to detect this autoimmune phenotype. This study will use these findings as a novel selection method of identifying long COVID patients with pathogenic IgG, thereby enriching the population most likely to benefit from immunoadsorption therapy.

This biomarker-guided personalized medicine approach could enhance treatment efficacy and advances long COVID therapeutic strategies. Additionally, the placebo-controlled and double blinded design will be needed to evaluate the true potential of autoantibodies adsorption therapy in long COVID. This study can add to our understanding on the role of autoantibodies in the pathogenesis of long COVID and could help in the development of precision-based immunotherapy for patients such as immunoadsorption.

ELIGIBILITY:
Inclusion Criteria:

* Long COVID based on the WHO-criteria
* PEM according to the DSQ-PEM
* BELL's functionality score 20-70%
* Good health prior to the long COVID diagnosis (WHO performance score 0)

Exclusion Criteria:

* Medical history of clinically significant respiratory- or cardiovascular disease
* Prior interventional cardiac procedure within 3 months prior to randomization
* Active immunosuppresive treatment for systemic autoimmune disorders
* Diabetes type 1
* Solid organ malignancy in the last 5 years
* Active psychiatric disorder currently under treatment by a psychiatrist
* BMI > 35
* Pre-existing fatigue
* Poor performance score prior to the long COVID diagnosis (WHO performance >0)
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-12 (Estimated); Study Completion 2028-03-12 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue measured by the Fatigue Assessment Scale (FAS) | At baseline and 28 days after start treatment
  Score range 10-50 (10 items, Likert scale 1-5). Higher scores indicate more severe fatigue (worse). The difference in scores from baseline will be measured (MCID of 4 points) as the primary outcome.

SECONDARY OUTCOMES:
Change in health related quality of life using the 36-Item Short Form Health Survey (SF-36) | At baseline and days 28, 60, 90, and 180
  Eight domains scored from 0-100. Domain scores are commonly summarized into the Physical Component Summary (PCS) and Mental Component Summary (MCS) (norm-based, mean 50, SD 10). Higher scores indicate better health-related quality of life and functioning.
Change in cognitive functioning using the Patient-Reported Outcomes Measurement Information System (PROMIS®) Cognitive Function Short Form 8a (PROMIS Cognitive Function Short Form 8a) | At baseline and days 28, 60, 90, and 180
  Raw scores are converted to T-scores (20-80), with a population mean of 50 (SD 10). Higher scores indicate better cognitive functioning. Change in score will be measured (MCID 3-5).
Change in autonomic symptoms using the Composite Autonomic Symptom Score-31 (COMPASS-31) | At baseline and days 28, 60, 90, and 180
  0-100 weighted total score across six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor symptoms. Higher scores indicate greater autonomic symptom burden.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) related to the intervention | From first study intervention through day 180
  All AEs and SAEs will be recorded, graded according to CTCAE v5.0, and assessed for relatedness to the study treatment. Specific attention will be given to complications of extracorporeal procedures (e.g., hypotension, bleeding, allergic reactions, infection, and vascular access issues)
Repeated Handgrip Strength | At baseline and days 28, 60, 90, and 180
  Handgrip strength will be assessed using a calibrated handheld dynamometer at four standardized measurement points in accordance with the American Society of Hand Therapists (ASHT) guidelines. Grip strength will be recorded in kilograms (kg). Higher grip strength reflects better muscle function.
Orthostatic intolerance using the NASA lean test | At baseline and days 28 and 180
  The NASA Lean Test is a standardized active standing test used to assess orthostatic intolerance. Participants rest in a supine position followed by an active standing phase while leaning against a wall to minimize skeletal muscle pumping. Heart rate and blood pressure are measured at predefined intervals during standing. Abnormal heart rate and/or blood pressure responses during the test indicate orthostatic intolerance.
Efficacy treatment by measuring immunoglobuline titers | At baseline (prior to treatment initiation), during treatment, and at days 28 and 180 after treatment initiation.
  Immunoglobulin G titers will be measured in blood samples using standardized laboratory assays and reported as concentrations (g/L).
Autoantibody score using an in-house Luminex assay | At screening and on days 28, 60, 90, and 180
  For this assay, IgG will be isolated from patient serum samples obtained during screening and analyzed using a Luminex-based multiplex immunoassay targeting a panel of 15 validated autoantigens. A weighted scoring system is applied to the resulting autoantibody signals.

CONTACTS AND LOCATIONS:
Locations (1):
- AUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
all request will be discussed within the study team